CLINICAL TRIAL: NCT02612038
Title: Nasal Expiratory Resistance in Patients With Sleep Apnea and Expiratory Flow Limitation
Acronym: ExpFLOSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding was available for the study
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012P000957E
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Expiratory flow limitation
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expiratory resistance (Experimental): Generic expiratory resistance will be added to the patient's respiratory circuit
  Interventions: Device: Expiratory resistance
- Sham expiratory resistance (Sham Comparator): Sham resistance will be added to the patient's respiratory circuit
  Interventions: Device: Sham expiratory resistance

INTERVENTIONS:
Device: Expiratory resistance — Generic expiratory resistance will be added to the patient's respiratory circuit
  Other Names: Expiratory positive pressure
  Arms: Expiratory resistance
Device: Sham expiratory resistance — Sham expiratory resistance will be added to the patient's respiratory circuit
  Arms: Sham expiratory resistance

SUMMARY:
Obstructive sleep apnea (OSA) is inherently site-specific. In a physiological controlled intervention study, the investigators seek to determine whether applying expiratory resistance can acutely improve ventilation and sleep in patients with expiratory flow limitation (EFL).

DETAILED DESCRIPTION:
Collapse of the upper airway can occur at different sites of the pharynx. One common and recognizable form of pharyngeal collapse is prolapse of the soft palate (velopharynx) on expiration, a phenomenon referred to as expiratory flow limitation (EFL). In principle, application of nasal positive expiratory pressure should reverse expiratory narrowing, increase ventilation, and prevent the subsequent progressive loss of airflow that leads to arousal from sleep, thereby improving OSA. One means to achieve this expiratory pressure is with the use of an added nasal expiratory resistance.

Accordingly, during a single night protocol, the investigators will examine the effects of increasing nasal expiratory resistance during sleep. During obstructed breathing, patients will be switched acutely, in random order, from normal conditions to an added expiratory resistance (30-80 cmH2O/L.s) or a sham resistance, for short (1 min) and prolonged periods (1 hour), repeatedly overnight.

Patients participating in the study will be divided into two groups, those exhibiting EFL versus those without EFL (i.e. with inspiratory flow limitation).

The main outcomes of the short physiologic interventions are:

* Increase in ventilation, and
* Increased time to a respiratory-related arousal from sleep, relative to sham conditions.

The main outcome of the prolonged interventions is:

--Reduced frequency of respiratory events (AHI; 3% desaturation or arousal) relative to sham conditions.

The central objective of the study is to test whether there is a greater improvement in the above outcomes in those with EFL versus those without EFL.

This data will allow us to test whether expiratory resistance is of potential therapeutic benefit specifically in patients with EFL rather than those without EFL.

ELIGIBILITY:
Inclusion Criteria:

* Presence of obstructive sleep apnea (AHI>10/hr)

Exclusion Criteria:

* Serious co-morbidities including lung disease, heart disease, renal disease
* Medications affecting respiration or sleep

Expiratory flow limitation (EFL) subgroup inclusion criteria: presence of clear EFL on polysomnographic study (reduced flow and increased pharyngeal pressure during expiration as a predominant cause of airflow obstruction).

non-EFL subgroup inclusion criteria: complete absence of EFL on polysomnographic study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Increase in ventilation (L/min) from baseline | Acutely (1 min)

SECONDARY OUTCOMES:
Increase in time to arousal from sleep | Acutely (1 min)
Reduction in frequency of respiratory events (apnea-hypopnea index, 3% desat/arousal; NREM supine) | Acutely (1 hour)

OTHER OUTCOMES:
Reduction in frequency of arousals from sleep | Acutely (1 hour)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wellman, PhD MD, Principal Investigator — Brigham and Women's Hospital